CLINICAL TRIAL: NCT06260280
Title: Relationship Between Chronic Sleep Deprivation and Changes in Cortical and Hippocampal Volume Assessed by Nuclear Magnetic Resonance in First-Year Medical Residents
Brief Title: Chronic Sleep Deprivation and Changes in Cortical and Hippocampal Volume
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Hilda Elizabeth Macías Cervantes, PhD, Instituto Mexicano del Seguro Social
Other Study IDs: 4
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Sleep Deprivation; Hippocampal Atrophy; Cortical Irregularity
Keywords: Sleep Deprivation; Hippocampal Atrophy; Cortical Irregularity; First-year medical residents
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First-year medical residents: All first-year residents entering our department for any of the different specialties will undergo a nuclear magnetic resonance scan before starting their shifts and a control scan 2 months into their residency to evaluate if there is an association between chronic sleep deprivation and changes in cortical and hippocampal volume.
  Interventions: Diagnostic Test: Cerebral Nuclear Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Cerebral Nuclear Magnetic Resonance — Cerebral Nuclear Magnetic Resonance before the start of the shifts and a control 2 months after the start of the residency to evaluate if there is an association between chronic sleep deprivation and changes in cortical and hippocampal volume.

SUMMARY:
Sleep is a physiological state that is essential for human performance, including academic, occupational, interpersonal, and psychological aspects. Sleep disruption or deprivation leads to a loss of psychomotor skills and an increased association with various diseases. Therefore, it is critical to assess how chronic sleep deprivation affects medical residents who work long shifts, including those assigned during their training.

DETAILED DESCRIPTION:
Objective: To determine if there is an association between chronic sleep deprivation and changes in cortical and hippocampal volume, assessed by nuclear magnetic resonance, in first-year medical residents assigned to the High Specialty Medical Unit, Specialty Hospital No. 1, National Medical Center of Bajío, during a period of 2 months after their admission.

Materials and Methods: This is a retrospective cohort study of first-year residents at UMAE T1, with a calculated sample size of 37 patients. Results are presented using descriptive statistics with mean and standard deviation or median with confidence intervals, depending on the type of variable. The relationship between MRI values and sleep deprivation will be assessed using Pearson's correlation coefficient or its non-parametric equivalent.

Ethical considerations: The study will be conducted with the informed consent of the patients in accordance with the General Health Law on Research and the Helsinki Declaration of 1975. The risk associated with this study is more than minimal.

Resources: Magnetic resonance studies will be performed at the High Specialty Medical Unit, Specialty Hospital No. 1, National Medical Center of Bajio, under the supervision of affiliated physicians specializing in the field of radiology and a fourth year resident in Diagnostic and Therapeutic Imaging.

ELIGIBILITY:
Inclusion Criteria:

* New resident physicians assigned to the High Specialty Medical Unit, Hospital de Especialidades No. 1 Centro Médico Nacional Del Bajío.

Exclusion Criteria:

* - Patients who have ingested caffeine, nicotine or alcohol in the last 24 hours.
* Patients with sleep disorders who present a score greater than 5 in the initial assessment of the Pittsburgh Sleep Quality Index.
* Patients with psychiatric treatment.
* Patients ingesting medications that intervene in the awake state.
* Patients with drug abuse (marijuana, cocaine, etc.).
* Patients with claustrophobia.
* Patients with metallic implants.

Ages: 24 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All first-year medical residents admitted to our hospital unit who meet the inclusion criteria will be informed of the purpose of the study and, after signing the informed consent, will undergo cranial magnetic resonance imaging.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2024-02-26 (Estimated); Primary Completion 2024-05-26 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hippocampal volumetry. | 2 months
  The hippocampal volume is obtained using the three planes of visualization of T1-weighted images in volumetric sequences. Volumetric analysis will be performed using volBrain and will be reported in cm3.
Change in cortical volumetry | 2 months
  The cortical volume is obtained using the three planes of visualization of T1-weighted images in volumetric sequences. Volumetric analysis will be performed using volBrain and will be reported in cm3.

CONTACTS AND LOCATIONS:
Overall Officials: Hilda E Macias, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Unidad Medica de Alta Especialidad No. 1, Bajío, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mason GM, Lokhandwala S, Riggins T, Spencer RMC. Sleep and human cognitive development. Sleep Med Rev. 2021 Jun;57:101472. doi: 10.1016/j.smrv.2021.101472. Epub 2021 Mar 13. PMID 33827030
- [Result] Craven J, McCartney D, Desbrow B, Sabapathy S, Bellinger P, Roberts L, Irwin C. Effects of Acute Sleep Loss on Physical Performance: A Systematic and Meta-Analytical Review. Sports Med. 2022 Nov;52(11):2669-2690. doi: 10.1007/s40279-022-01706-y. Epub 2022 Jun 16. PMID 35708888
- [Result] Perotta B, Arantes-Costa FM, Enns SC, Figueiro-Filho EA, Paro H, Santos IS, Lorenzi-Filho G, Martins MA, Tempski PZ. Sleepiness, sleep deprivation, quality of life, mental symptoms and perception of academic environment in medical students. BMC Med Educ. 2021 Feb 17;21(1):111. doi: 10.1186/s12909-021-02544-8. PMID 33596885
- [Result] Baumann Q, Bulaid Y, Van Vliet A, Gabrion A, Klein C, Mertl P. Sleep Deprivation Adversely Impacts Resident Performance for Simulated Arthroscopy. Arthrosc Sports Med Rehabil. 2021 Jul 9;3(4):e1125-e1132. doi: 10.1016/j.asmr.2021.04.001. eCollection 2021 Aug. PMID 34430893
- [Result] Dai XJ, Jiang J, Zhang Z, Nie X, Liu BX, Pei L, Gong H, Hu J, Lu G, Zhan Y. Plasticity and Susceptibility of Brain Morphometry Alterations to Insufficient Sleep. Front Psychiatry. 2018 Jun 27;9:266. doi: 10.3389/fpsyt.2018.00266. eCollection 2018. PMID 29997530
- [Result] Elvsashagen T, Zak N, Norbom LB, Pedersen PO, Quraishi SH, Bjornerud A, Alnaes D, Doan NT, Malt UF, Groote IR, Westlye LT. Evidence for cortical structural plasticity in humans after a day of waking and sleep deprivation. Neuroimage. 2017 Aug 1;156:214-223. doi: 10.1016/j.neuroimage.2017.05.027. Epub 2017 May 17. PMID 28526620